CLINICAL TRIAL: NCT05333913
Title: Prevalence of Functional Iron Deficiency (FID) and Quality of Life (QoL) in Patients with Oncological and with Haematological Malignancies
Brief Title: Prevalence of FID and QoL in Patients with Oncological and with Haematological Malignancies
Status: Completed | Type: Observational
Sponsor: Luzerner Kantonsspital (Other)
Responsible Party: Principal Investigator, Axel Rüfer, MD, Co-Head Physician, Luzerner Kantonsspital
Other Study IDs: Kantonsspital_Luzern
Record Dates: First submitted 2022-04-11; First posted 2022-04-19 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2022-04

CONDITIONS: Functional Iron Deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Prospective single-center observational study assessing prevalence of FID (Laboratory work-up) and Quality of Life (Questionnaire) in adult patients with oncological and with haematological malignancies within four weeks prior to disease-directed therapy.

DETAILED DESCRIPTION:
Patients included into the study will have a laboratory work-up assessing the occurence of functional iron deficiency using laboratory parameters (full blood count, reticulocytes, transferrin saturation, serum-ferritin, CRP, ALAT) and have to fill in once the FACT-An questionnaire generating data on Quality of Life at time of study entry.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Patients with oncological (solid tumors) and with haematological malignancies (non-solid tumors, including Plasma cell myeloma, lymphoma, myeloproliferative neoplasias [MPN], myelodysplastic syndromes [MDS] and chronic leukemias)
* Within four weeks prior to disease-directed systemic therapy
* Participation in other trials is possible

Exclusion Criteria:

* Known iron deficiency with or without iron substitution p.o. or i.v. within last 8 weeks prior to inclusion into this trial
* Therapy with RBC-transfusions within last 8 weeks prior to inclusion into this trial
* Therapy with ESA within last 8 weeks prior to inclusion into this trial
* Malignancies with acute need for therapeutic intervention (e.g. acute leukemias, superior vena cava obstruction, etc.)
* Pregnancy
* Any other serious underlying medical, psychiatric, psychological, familial or geographical condition, which in the judgment of the investigator may interfere with the trial
* Inability to give consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with oncological (solid tumors) and with haematological malignancies (non-solid tumors, including Plasma cell myeloma, lymphoma, myeloproliferative neoplasias [MPN], myelodysplastic syndromes [MDS] and chronic leukemias)
  Study entry within four weeks prior to disease-directed systemic therapy
Sampling Method: Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2022-02-07 (Actual); Primary Completion 2023-04-04 (Actual); Study Completion 2023-04-04 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is the determination of the prevalence of FID in patients with oncological and with haematological malignancies. | through study completion, an average of 1 year
  Prevalence of functional iron deficiency in the study population using full blood count, reticulocytes, transferrin saturation, serum-ferritin, CRP and ALAT.

SECONDARY OUTCOMES:
The secondary endpoint is the collection of data on quality of life using FACT-An. | through study completion, an average of 1 year
  Data on quality of life using FACT-An, which covers a fatigue and anemia subscale, as well as generic QoL domains including physical well-being, functional well-being, emotional well-being and socal well-being subscales - this is done at study entry estimating scores at various subscales of FACT-An.

CONTACTS AND LOCATIONS:
Overall Officials: Axel Ruefer, MD, Study Chair — Hematology Department, Luzerner Kantonsspital, 6000 Luzern 16, Switzerland
Locations (1):
- Luzerner Kantonsspital, Lucerne, Canton of Lucerne, Switzerland

IPD SHARING:
Plan to Share IPD: No